CLINICAL TRIAL: NCT02364440
Title: Safety and Efficacy Evaluation of Ultherapy™ System in Aging Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: E-1405/250-001
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-02

CONDITIONS: Wrinkles
Keywords: skin laxity; Ultherapy™ System; rhytids
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy™ System (Experimental): Ultherapy™ System
  Interventions: Device: Ultherapy™ System

INTERVENTIONS:
Device: Ultherapy™ System — Subjects will receive 20 lines Ultherapy™ System Treatment over their right and left hand with 1.5 and 3.0 probe respectively

SUMMARY:
Enrolled subjects will receive Ultherapy™ System treatment on the back of their both hands. Follow-up visits will occur at 90 days post-treatment. Study photos will be obtained pre-treatment and at 90 days post-treatment

DETAILED DESCRIPTION:
Before Treatment:

The subject's eligibility (inclusion/exclusion criteria) will be assessed, and the 5-point Hand Grading Scale wil be evaluated by the Investigator in charge of assessment.

Treatment:

The Investigator will apply to the eligible subject the Study Device Ultherapy™ System with 20 lines of 1.5 and 3.0 probe respectively to the back of the left and right hand .

Post-Treatment:

All subjects will visit the Institution at12 weeks from the day of procedure, and will take photos of the back of the hands. Efficacy evaluation will performed by the Photographic Evaluator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years.
* Score of 1 to 3 on The 5-point Hand Grading Scale
* Subjects who understand the study contents and signed the informed consent

Exclusion Criteria:

* Presence of an active systemic infectious disease
* Significant scarring in the hand to be treated
* Previous episode of surgery in the hand to be treated
* Subjects who have aesthetic addiction, drug abuse, alcohol abuse

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Investigator's evaluation of 5-point Hand grading scale | 12 weeks post-treatment
  2 assessors will be evaluate 5-point Hand grading scale from baseline and 12weeks post treatment

SECONDARY OUTCOMES:
Subject Assessment of Improvement at 12 weeks post-treatment | 12 weeks post-treatment
  Subjects complete a Patient Assessment Global Aesthetic Improvement Scale at 12 weeks post-treatment
Investigator Assessment of Improvement at 12 weeks post-treatment | 12 weeks post-treatment
  Investigator complete Global Aesthetic Improvement Scale at 12 weeks post-treatment by comparing subject's photographs
Subjects' Assessment of Pain during treatment | Subjects were assessed for the duration of study treatment
  Pain score record using a Numeric Rating Scale (NRS,0-10) , with 0 representing no pain and 10 representing the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: ChangSik Pak, Bachelor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea